CLINICAL TRIAL: NCT05039840
Title: Efficacy and Safety of SAR441344 in the Treatment of Systemic Lupus Erythematosus: A Randomized, Double Blind, Placebo-controlled, Phase 2, Proof of Concept Study
Brief Title: Efficacy and Safety of Frexalimab (SAR441344) in the Treatment of Systemic Lupus Erythematosus
Acronym: APATURA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17010; U1111-1266-5011 (Registry Identifier: ICTRP); 2023-508654-26 (Registry Identifier: CTIS); 2021-001567-25 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Frexalimab (Experimental): Frexalimab intravenous (IV) loading dose followed by subcutaneous (SC) doses, 24 weeks
  Interventions: Drug: SAR441344 IV; Drug: SAR441344 SC
- Placebo (Placebo Comparator): Placebo IV loading dose followed by SC, 24 weeks
  Interventions: Drug: Placebo IV; Drug: Placebo SC

INTERVENTIONS:
Drug: SAR441344 IV — Pharmaceutical form: solution Route of administration: Intravenous infusion
  Arms: Frexalimab
Drug: SAR441344 SC — Pharmaceutical form: solution Route of administration: subcutaneous injection
  Arms: Frexalimab
Drug: Placebo IV — Pharmaceutical form: solution Route of administration: Intravenous infusion
  Arms: Placebo
Drug: Placebo SC — Pharmaceutical form: solution Route of administration: subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multinational, randomized, placebo-controlled, parallel treatment, Phase 2, double-blind, 2 arm study evaluating the efficacy and safety of SAR441344 in comparison with placebo in the treatment of participants aged 18 to 70 years with active Systemic Lupus Erythematosus (SLE). Study details include:

* Study duration: 36 weeks
* Treatment duration: 24 weeks
* Visit frequency: every 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE for at least 6 months prior to screening by fulfilling the Revised Criteria for Classification of SLE according to the 1997 Update of the 1982 ACR criteria
* Positive antinuclear antibody (ANA) (titer ≥1:80) during screening
* Positivity for at least one serological characteristic
* Total hSELENA-SLEDAI score ≥6 (including points attributed from arthritis and rash) during screening and at least 4 points from clinical features at randomization as confirmed by a Sponsor-selected independent reviewer(s)
* At least 1 BILAG A score or 2 BILAG B scores during screening as confirmed by a Sponsor-selected independent reviewer(s)
* Receiving at least one of the standard of care (SOC) for SLE (combination is possible)
* Body weight within 45 kg to 120 kg (inclusive) at screening
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Primary diagnosis of a rheumatic disease besides SLE or an inflammatory joint or skin disease other than SLE that could confound the disease activity assessments
* Active and severe lupus nephritis
* Active severe or unstable neuropsychiatric SLE including but not limited to seizures, psychosis, acute confusional state, transverse myelitis, central nervous system vasculitis and optic neuritis
* Known or suspected drug-induced lupus
* History, clinical evidence, suspicion or significant risk, for thromboembolic events, as well as myocardial infarction, stroke, and/or antiphospholipid syndrome and any participants requiring antithrombotic treatment
* History or current hypogammaglobulinemia
* Serious systemic viral, bacterial or fungal infection
* Participants with a history of invasive opportunistic infections, such as, but not limited to histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumocystis jirovecii, and aspergillosis, regardless of resolution
* Evidence of active or untreated latent tuberculosis as documented by medical history (eg, chest Xrays) and examination, and tuberculosis testing
* High dose of steroids, or a change in dose within 4 weeks prior to randomization
* High dose of antimalarial, or a change in dose within 12 weeks prior to randomization
* High dose of immunosuppressants or a change in dose within 12 weeks prior to randomization
* Use of cyclophosphamide within 3 months prior to screening
* Previous parenteral (IV), intramuscular (IM), or intra-articular steroid administration within 4 weeks prior to randomization
* Participants likely to require multiple courses of oral corticosteroid (OCS) during the study for chronic diseases other than SLE
* Administration of any live (attenuated) vaccine within 3 months prior to randomization (eg, varicella zoster vaccine, oral polio, rabies)
* Administration of any non-live vaccine (eg, seasonal influenza, COVID-19) within 4 weeks prior to randomization

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieved a Systemic Lupus Erythematosus Responder Index (SRI-4) response at Week 24. | At Week 24
  A composite endpoint, with SRI-4 response requiring a ≥ 4-point improvement (reduction) from baseline in Hybrid Safety of Estrogens in Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (hSELENA-SLEDAI), no new British Isles Lupus Assessment Group (BILAG-2004) A organ domain scores, or ≥ 2 new BILAG-2004 B organ domain scores compared with baseline, no worsening from baseline in lupus disease activity, and no permanent discontinuation of study drug or use of new or increased medication for SLE other than defined per protocol.

SECONDARY OUTCOMES:
Percentage of participants who achieved an SRI-4 response in prespecified biomarker (BM) subgroups at Week 24 | At Week 24
Percentage of participants who achieved a BILAG-based Composite Lupus Assessment (BICLA) response in prespecified BM subgroups at Week 24 | At Week 24
Percentage of participants who achieved a BICLA response at Week 24 | At Week 24
Percentage of participants whose prednisone dose was ≤ 7.5 mg at Week 16 and maintained through Week 24 in the subgroup with baseline prednisone ≥10 mg/day | Until Week 24
Total cumulative corticosteroid dose over 24 weeks | Until Week 24
Percentage of participants achieving an SRI-4 response at week 24 with sustained reduction of oral corticosteroids | At Week 24
Percent change from baseline in percentage in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI)-A at Week 24 in the subgroup of participants with baseline CLASI-A score ≥8 | At Week 24
Percentage of participants with ≥50% improvement in CLASI-A at Week 24 in the subgroup of participants with baseline CLASI-A score ≥8 | At Week 24
Percentage of participants with ≥50% improvement in the number of tender and swollen joints at Week 24 (among participants with at least 4 joints affected at baseline) | At Week 24
Incidence of treatment-emergent AEs (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs) from Baseline to Week 36 End of Study (EoS) | Until Week 36
Incidence of study investigational medicinal product permanent discontinuations and study withdrawals due to TEAEs from Baseline to Week 36 (EoS) | Until Week 36
Participants with medically significant changes in vital signs, electrocardiogram (ECG), and/or laboratory evaluation | Until Week 36
Measurement of anti-drug antibodies (ADA) (before administration at Week 0, 4, 8, 12, 16, 20, 24 and after treatment discontinuation at Week 36) | Until Week 36
SAR441344 concentrations over time | Until Week 36
Pharmacokinetic parameters: maximum concentration (Cmax) | Until Week 36
Pharmacokinetic parameters: time to Cmax (tmax) | Until Week 36
Pharmacokinetic parameters: area under the curve over the dosing interval (AUC0-tau) | Until Week 36
Pharmacokinetic parameters: terminal half-life (t1/2z). | Until Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (74):
- United States (22):
  - Accel Research Sites Network - Vestavia Hills- Site Number : 8400003, Vestavia Hills, Alabama
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Chandler- Site Number : 8400026, Chandler, Arizona
  - Arizona Arthritis & Rheumatology Associates - South Vineyard Avenue- Site Number : 8400022, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research - Sun City- Site Number : 8400027, Sun City, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson Southeast- Site Number : 8400023, Tucson, Arizona
  - Saint John's Physician Partners- Site Number : 8400015, Santa Monica, California
  - Millennium Clinical Trials - Simi Valley- Site Number : 8400004, Simi Valley, California
  - Omega Research Consultants - Debary - North Charles Richard Beall Boulevard- Site Number : 8400002, DeBary, Florida
  - Vitalia Medical Research - Margate- Site Number : 8400039, Margate, Florida
  - Innovia Research Center- Site Number : 8400037, Miramar, Florida
  - Integral Rheumatology and Immunology Specialists- Site Number : 8400014, Plantation, Florida
  - Infigo Clinical Research- Site Number : 8400016, Sanford, Florida
  - Inspire Santa Fe Medical Group- Site Number : 8400019, Santa Fe, New Mexico
  - Columbia University Irving Medical Center- Site Number : 8400009, New York, New York
  - RAO - Rheumatology Associates of Oklahoma- Site Number : 8400013, Oklahoma City, Oklahoma
  - Private Practice - Dr. Ramesh C. Gupta I- Site Number : 8400008, Memphis, Tennessee
  - Tekton Research - West Gate- Site Number : 8400001, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions - Colleyville- Site Number : 8400017, Colleyville, Texas
  - Lone Start Arthritis & Rheumatology Associates- Site Number : 8400025, Fort Worth, Texas
  - Prolato Clinical Research Center- Site Number : 8400005, Houston, Texas
  - AARA Clinical Research - Lone Star Arthritis & Rheumatology Associates - Irving- Site Number : 8400024, Irving, Texas
  - West Texas Clinical Research- Site Number : 8400018, Lubbock, Texas
- Argentina (6):
  - Investigational Site Number : 0320008, Berazategui, Buenos Aires
  - Investigational Site Number : 0320003, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
- Brazil (5):
  - Centro de Estudos em Terapias Inovadoras- Site Number : 0760002, Curitiba, Paraná
  - LMK Servicos Medicos- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto- Site Number : 0760006, São José do Rio Preto, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino- Site Number : 0760007, São Paulo
  - Centro Paulista de Investigaçăo Clínica - CEPIC- Site Number : 0760004, São Paulo
- Chile (4):
  - Investigational Site Number : 1520002, Osorno, Los Lagos Region
  - Investigational Site Number : 1520003, Talca, Maule Region
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- Georgia (5):
  - Investigational Site Number : 2680005, Tbilisi
  - Investigational Site Number : 2680004, Tbilisi
  - Investigational Site Number : 2680001, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680002, Tbilisi
- Greece (5):
  - Investigational Site Number : 3000004, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Heraklion
  - Investigational Site Number : 3000005, Larissa
  - Investigational Site Number : 3000002, Thessaloniki
- Hungary (2):
  - Investigational Site Number : 3480002, Gyula
  - Investigational Site Number : 3480003, Székesfehérvár
- Italy (3):
  - IRCCS Ospedale San Raffaele-Site Number : 3800001, Milan, Milano
  - Investigational Site Number: 3800004, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli-Site Number : 3800002, Rome, Roma
- Investigational Site Number : 4800001, Vacoas, Mauritius
- Mexico (8):
  - Investigational Site Number : 4840009, Mexico City, Mexico City
  - Investigational Site Number : 4840004, Mexico City, Mexico City
  - Investigational Site Number : 4840001, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, Mérida, Yucatán
  - Investigational Site Number : 4840006, Chihuahua City
  - Investigational Site Number : 4840011, Chihuahua City
  - Investigational Site Number : 4840007, Mexico City
  - Investigational Site Number : 4840008, Veracruz
- GCM Medical Group - San Juan - Calle Jose Marti- Site Number : 8400011, San Juan, Puerto Rico
- Investigational Site Number : 6430002, Moscow, Russia
- Spain (4):
  - Investigational Site Number : 7240002, Sabadell, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240005, Valencia
  - Investigational Site Number : 7240004, Valladolid
- Investigational Site Number : 7560001, Sankt Gallen, Switzerland
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920003, Ankara
  - Investigational Site Number : 7920002, Denizli
  - Investigational Site Number : 7920004, Sakarya
- Ukraine (3):
  - Investigational Site Number : 8040006, Kyiv
  - Investigational Site Number : 8040001, Kyiv
  - Investigational Site Number : 8040005, Poltava

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- See also: ACT17010 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25207&tenant=MT_SNY_9011